CLINICAL TRIAL: NCT04034485
Title: Randomized, Open-Label, Cross-Over, Phase 3 Study to Evaluate the Efficacy and Safety of LIB003 With Evolocumab in Homozygous Familial Hypercholesterolemia Patients on Stable Lipid-Lowering Therapy
Brief Title: Phase 3 Study to Evaluate the Efficacy and Safety of LIB003 With Evolocumab in HoFH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LIB Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LIB003-003
Record Dates: First submitted 2019-07-22; First posted 2019-07-26 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Homozygous Familial Hypercholesterolemia
Keywords: LDL cholesterol; PCSK9 inhibition
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia | interventions — evolocumab

STUDY DESIGN:
Intervention Model Description: open label, randomized, cross-over
Masking Description: treatment is open label but lipid results are masked to participant, investigator and sponsor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LIB003 (lerodalcibep) (Experimental): 300 mg SC Q4W
  Interventions: Drug: lerodalcibep
- evolocumab (Active Comparator): 420 mg SC Q4W
  Interventions: Drug: evolocumab

INTERVENTIONS:
Drug: lerodalcibep — PCSK9 inhibitor
  Other Names: LIB003
  Arms: LIB003 (lerodalcibep)
Drug: evolocumab — PCSK9 inhibitor
  Other Names: Repatha
  Arms: evolocumab

SUMMARY:
To compare the safety, tolerability and LDL-C response after 24 Weeks of monthly (every 4 weeks [Q4W]) subcutaneous (SC) dosing of LIB003 300 mg with monthly (Q4W) SC dosing of 420 mg evolocumab (Repatha®) in patients with HoFH on stable diet and oral LDL-C-lowering drug therapy

DETAILED DESCRIPTION:
Patients with verified HoFH on stable and continuing doses of oral lipid lowering therapy will be randomized to either evolocumab 420 mg Q4W or LIB003 300 mg Q4W for 24 weeks (Period A). At Week 24, subjects will be crossed over to LIB003 if they were on evolocumab and vice versa for the next 24 weeks (Period B).

ELIGIBILITY:
Inclusion Criteria:

* HoFH diagnosed clinically and confirmed by genotyping
* Weight of >30 kg and body mass index (BMI) >17 and <40 kg/m2
* stable diet and lipid-lowering oral therapies for at least 4 weeks

Exclusion Criteria:

* mipomersen within 6 months of screening;
* LDL or plasma apheresis <2 months prior to randomization
* history of non-response to PCSK9 mAb or presence of receptor negative/null LDLR activity expected to result in non-response to PCSK9 inhibition
* prior or active clinical condition or acute and/or unstable systemic disease compromising subject inclusion

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-12-07 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Percent reduction in Low Density Lipoprotein Cholesterol (LDL-C) at week 24 | baseline to 24 weeks on each treatment
  Change in serum LDL-C from baseline after 24 weeks

SECONDARY OUTCOMES:
The incidence and severity of treatment emergent adverse events (TEAEs) | baseline to 24 weeks on each treatment
  safety and tolerability will be based on the incidence and severity of treatment emergent adverse events

OTHER OUTCOMES:
Percent reduction in lipoprotein (a) [Lp(a)] at week 24 | baseline to 24 weeks on each treatment
  Change in serum Lp(a) from baseline after 24 weeks
Percent reduction in apolipoprotein B (Apo B) at week 24 | baseline to 24 weeks on each treatment
  Change in serum Apo B from baseline after 24 weeks
Presence of anti LIB003 antibodies (ADAs) | baseline to 24 weeks
  Measurement of ADAs at baseline and various intervals

CONTACTS AND LOCATIONS:
Overall Officials: Evan A Stein, MD PhD, Study Director — LIB Therapeutics
Locations (12):
- United States (2):
  - NorthShore University Health System, Evanston, Illinois
  - Metabolic & Atherosclerosis Research Center (MARC), Cincinnati, Ohio
- India (3):
  - VMMC & Safdarjung Hospital, Delhi, National Capital Territory of Delhi
  - CIMS Hospital Pvt. Ltd, Ahmedabad
  - G.B. Pant Institute of Postgraduate Medical Education & Research, New Delhi
- Israel (2):
  - Department of Medicine, Hadassah University Hospital, Jerusalem
  - Rabin Medical Center, Beilinson Hospital,, Petah Tikva
- Lipid Clinic, Oslo University Hospital, Oslo, Norway
- South Africa (2):
  - Carbohydrate and Lipid Metabolism Research Unit, Johannesburg, Gauteng
  - Division of Lipidology, Department of Medicine University of Cape Town, Cape Town, Western Province
- Turkey (Türkiye) (2):
  - Ege University Medical School, Izmir, Bornova
  - Afyonkarahisar Health Sciences University, Afyonkarahisar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raal FJ, Mehta V, Kayikcioglu M, Blom D, Gupta P, Elis A, Turner T, Daniels C, Vest J, Mitchell T, Caldwell K, Bahassi EM, Kallend D, Stein EA. Lerodalcibep and evolocumab for the treatment of homozygous familial hypercholesterolaemia with PCSK9 inhibition (LIBerate-HoFH): a phase 3, randomised, open-label, crossover, non-inferiority trial. Lancet Diabetes Endocrinol. 2025 Mar;13(3):178-187. doi: 10.1016/S2213-8587(24)00313-9. Epub 2025 Jan 24. PMID 39870096